CLINICAL TRIAL: NCT06642571
Title: Investigation of Pharmacokinetics of 2 Different Formulations of NNC0519-0130 in Adult Participants With Overweight or Obesity
Brief Title: A Research Study to Compare How Much of the Medicine NNC0519-0130 is in the Blood of People With Overweight or Obesity Who Receive 2 Preparations of the Medicine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9541-4919; U1111-1307-3788 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1a: NNC0519-0130 C and NNC0519-0130 B (Experimental): Participants will start treatment with formulation NNC0519-0130 C and receive a pre-determined dose escalation regimen of NNC0519-0130 B and NNC0519-0130 C.
  Interventions: Drug: NNC0519-0130 B; Drug: NNC0519-0130 C
- Part 1b: NNC0519-0130 B and NNC0519-0130 C (Experimental): Participants will start treatment with formulation NNC0519-0130 B and receive a pre-determined dose escalation regimen of NNC0519-0130 B and NNC0519-0130 C.
  Interventions: Drug: NNC0519-0130 B; Drug: NNC0519-0130 C
- Part 2a: NNC0519-0130 B and NNC0519-0130 C (Experimental): Participants will receive a pre-determined dose escalation regimen of NNC0519-0130 B in run-in period followed by treatment with NNC0519-0130 B then NNC0519-0130 C.
  Interventions: Drug: NNC0519-0130 B; Drug: NNC0519-0130 C
- Part 2b: NNC0519-0130 C and NNC0519-0130 B (Experimental): Participants will receive a pre-determined dose escalation regimen of NNC0519-0130 B in run-in period followed by treatment with NNC0519-0130 C then NNC0519-0130 B.
  Interventions: Drug: NNC0519-0130 B; Drug: NNC0519-0130 C

INTERVENTIONS:
Drug: NNC0519-0130 B — NNC0519-0130 B will be administered subcutaneously.
Drug: NNC0519-0130 C — NNC0519-0130 C will be administered subcutaneously.

SUMMARY:
This study will look into a new study medicine called NNC0519-0130 to improve the treatment option for people living with excess body weight or type 2 diabetes or both. The purpose of this study is to compare the amount of NNC0519-0130 in the blood of participants who have excess body weight. The study comprises two parts and the participants will receive both preparations NNC0519-0130 B and NNC0519-0130 C, which treatment the participants get is decided by chance. The study will last for about 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential.
* Age 18-64 years (both inclusive) at the time of signing the informed consent.
* Body Mass Index (BMI) between 27.0 kilogram per square meter (kg/m^2) and 39.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any condition which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Glycated hemoglobin (HbA1c) greater than or equal to (≥) 6.5 % (48 millimoles per mole [mmol/mol]) at screening.
* Use of prescription medicinal products or nonprescription drugs, except routine vitamins, occasional use of acetaminophen, ibuprofen, acetylsalicylic acid, or topical medication (including eye drops for pupil dilation) not reaching systemic circulation, within 14 days before screening.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
AUC,NNC0519-0130,SS: Area under the NNC0519-0130 plasma concentration-time curve during a dosing interval at steady state (SS) | From pre-dose up to 7 days post-dose
  Measured in hours*nanomoles per liter (h*nmol/L).

SECONDARY OUTCOMES:
Cmax,NNC0519-0130,SS: Maximum plasma concentration of NNC0519-0130 at steady state | From pre-dose up to 7 days post-dose
  Measured in nanomoles per liter (nmol/L).
Number of adverse events | From time of first dosing (day 1) until completion of the end of study visit (day 141/162)
  Measured in number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- ICON, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com